CLINICAL TRIAL: NCT02939209
Title: Preventing Rebound Pain After Arthroscopic Rotator Cuff Repair and/or Acromioplasty Under General Anesthesia and Interscalene Block: A Randomized Controlled Trial of Pre-emptive Opioid Treatment Compared to Placebo
Brief Title: Pre-emptive Opioid Treatment to Prevent Rebound Pain After Arthroscopic Rotator Cuff Repair and/or Acromioplasty Under General Anesthesia and Interscalene Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vishal Uppal (Other)
Responsible Party: Sponsor-Investigator, Vishal Uppal, Assistant Professor & Staff Anesthesiologist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1021783
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Rotator Cuff Injury; Pain
Keywords: Rotator cuff repair; Interscalene block; Hydromorphone; Pain; Rebound pain; Acromioplasty
MeSH Terms: conditions — Rotator Cuff Injuries; Pain | interventions — Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydromorphone (Experimental): Patients will be given 2 mg hydromorphone (immediate release) in the post anesthetic care unit.
  Interventions: Drug: Hydromorphone Hcl 2Mg Tab
- Placebo (Placebo Comparator): Patients will be given placebo in the post anesthetic care unit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydromorphone Hcl 2Mg Tab — Patients will be given 2 mg hydromorphone (immediate release formulation) in the post anesthetic care unit.
  Arms: Hydromorphone
Drug: Placebo — Patients may be randomized to placebo.
  Arms: Placebo

SUMMARY:
Arthroscopic shoulder rotator cuff repair and acromioplasty are associated with severe postoperative pain. The interscalene block (ISB) is commonly used for this type of surgery, providing analgesia by anesthetizing the nerves that supply the shoulder. Although the nerve block provides extremely effective analgesia for the first 6-8 hours, patients experience severe pain once its effect has regressed. This study will assess whether a single dose of oral hydromorphone controlled release, given to overlap the waning of the ISB, will improve postoperative pain control and reduce the incidence of rebound pain.

Seventy patients undergoing rotator cuff repair will receive standardized ISB and general anesthesia for the surgery. Six hours (+/- 1 hour) after ISB, the patients will randomly receive either a single oral dose of 2 mg Hydromorphone (immediate release formulation) or placebo. The patient will be then discharged home with a prescription for multimodal analgesia, which is the standard of care. Patients will be given a diary to record their pain scores and track use of analgesic medications for 24 hours. Twenty-four hours after the ISB, the patients will receive a phone call from a nurse as per the standard of care. During this phone call, questions will be asked about their pain control.

If a single dose of pre-emptive hydromorphone is demonstrated to be safe and effective, it will lead to change in practice of how we manage pain after rotator cuff repair. Furthermore, the finding of this study may apply to similar surgical procedures (such as elbow, knee and ankle repairs) that are associated with rebound pain when the nerve block wears off.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* scheduled to receive ISB and general anesthesia as a day surgery patient for rotator cuff repair and acromioplasty, as a part of planned routine care

Exclusion Criteria:

* Allergy, sensitivity, or absolute contraindications to any of the medications involved in the study
* preexisting CNS depression, or taking regularly medication that cause CNS depression
* preexisting cognitive deficits, dementia, or delirium
* severe respiratory comorbidities (e.g. chronic obstructive pulmonary disease, pneumonia, respiratory failure)
* sleep disordered breathing (diagnosed OSA, obesity hypoventilation syndrome)
* pregnancy and breast feeding
* history of chronic pain or regular (at least once daily) opioid use preoperatively
* renal impairment - CrCl ≤60 mL/minute
* not fluent in English to be able to participate in the study process, including consent and phone interview
* Body Mass Index >35
* inability to take oral medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Worst pain score | 24 hours post interscalene block
  We will investigate whether a single dose of hydromorphone 2 mg, given at six hours after single-shot ISB for rotator cuff repair, reduces worst pain score (NRS) in first 24 hours by two points or more as measured on 11 point (0-10) NRS scale when compared to placebo, with perioperative multimodal analgesia used in both groups.

SECONDARY OUTCOMES:
Time to first rescue opioid use, within 24 hours after ISB insertion | 24 hours post interscalene block
Total rescue hydromorphone consumption, within 24 hours after ISB insertion | 24 hours post interscalene block
Two hourly pain score (burden of pain) while the patient is awake | 24 hours post interscalene block
Incidence of clinically significant nausea and vomiting after the dose of study drug | 24 hours post interscalene block
Number of patients failing discharge from hospital due to pain, nausea, vomiting or sedation | 24 hours post interscalene block
Number of patients needing emergency room visit due to pain within 24 hours of surgery | 24 hours post interscalene block
Number of patients needing hospital readmission due to pain within 24 hours of surgery | 24 hours post interscalene block

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Uppal, Principal Investigator — Dalhousie Anesthesia
Locations (2):
- Canada (2):
  - Nova Scotia Health Authority Queen Elizabeth II Hospital Halifax Infirmary site, Halifax, Nova Scotia
  - St Joseph's (McMaster University), Hamilton, Ontario

REFERENCES:
- [Derived] Uppal V, Barry G, Ke JXC, Kwofie MK, Trenholm A, Khan M, Shephard A, Retter S, Shanthanna H. Reducing rebound pain severity after arthroscopic shoulder surgery under general anesthesia and interscalene block: a two-centre randomized controlled trial of pre-emptive opioid treatment compared with placebo. Can J Anaesth. 2024 Jun;71(6):773-783. doi: 10.1007/s12630-023-02594-0. Epub 2023 Oct 13. PMID 37833472